CLINICAL TRIAL: NCT00152269
Title: A Phase III, 12-Month, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety (Including Bone Density Assessment) of Two Doses of J867 Versus Placebo in Subjects With Uterine Leiomyomata
Brief Title: Treatment of Uterine Fibroids With Asoprisnil(J867)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M01-390
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Leiomyoma; Menorrhagia; Metrorrhagia
Keywords: Symptomatic Uterine Fibroids; Excessive Uterine Bleeding; Uterine Hemorrhage; asoprisnil
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Hemorrhage | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asoprisnil — 10mg Tablet, oral Daily for 12 months
  Arms: 1
Drug: Asoprisnil — 25mg Tablet, oral Daily for 12 months
  Arms: 2
Drug: Placebo — Placebo, Tablet, oral Daily for 12 months
  Arms: 3

SUMMARY:
The objective of this study is to determine the safety and effectiveness of asoprisnil in symptomatic women with abnormal uterine bleeding associated with uterine fibroids.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of abnormal uterine bleeding associated with uterine fibroids in women and many women must resort to surgery for relief. The objective of this study is to determine the safety and efficacy of asoprisnil 10 mg and 25 mg tablets, compared to placebo, administered daily for 12 months to women with abnormal uterine bleeding associated with uterine fibroids, by assessing whether asoprisnil administration prevents surgical and/or invasive intervention in the study population. Women, who meet the predefined uterine bleeding criteria for surgical and/or invasive intervention (hysterectomy, myomectomy, uterine artery embolization) who are willing to undergo surgical and/or invasive intervention if the study medication fails, will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* History of regular menstrual cycles (21-42 days)
* Diagnosis of uterine fibroid(s)
* Abnormal vaginal bleeding associated with uterine fibroids
* Otherwise in good health
* Agrees to undergo surgery (hysterectomy) or any other invasive procedure if the study medication fails
* Negative pregnancy test
* Agrees to Double-barrier method of contraception
* Pap smear with no evidence of malignancy or pre-malignant changes
* Endometrial biopsy with no significant histological disorder

Exclusion Criteria:

* Any abnormal lab or procedure result the study-doctor considers important
* Severe reaction(s) to or are currently using any hormone therapy
* History of osteoporosis or other bone disease
* Previous myomectomy with 1 year and/or previous uterine artery embolization within 6 months
* History of Polycystic Ovary Syndrome or prolactinoma
* MRI shows significant gynecologic disorder
* Uterine size > 25 weeks gestation
* Hemoglobin < 8 g/dL at Day -1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2002-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
The percent of subjects who demonstrate a clinically meaningful improvement in bleeding and do not have surgical/invasive intervention. | Month 12 or Final Visit

SECONDARY OUTCOMES:
Percent of subjects with clinically meaningful improvement in bleeding and who do not require surgical/invasive intervention. | Month 6
Change from baseline in menstrual pictogram score. | Final Month
Change from baseline in number of days with bleeding. | Final Month
Change from baseline in hemoglobin concentration. | Final Visit
Percent change from baseline in volume of the largest fibroid. | Final Visit
Change from baseline in bloating, pelvic pressure, dysmenorrhea and urinary symptoms. | Final Visit
Change from baseline in total symptom severity score and UFS-QOL total score. | Final Visit
Cumulative percent of subjects who achieve amenorrhea. | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott

REFERENCES:
- [Derived] Stewart EA, Diamond MP, Williams ARW, Carr BR, Myers ER, Feldman RA, Elger W, Mattia-Goldberg C, Schwefel BM, Chwalisz K. Safety and efficacy of the selective progesterone receptor modulator asoprisnil for heavy menstrual bleeding with uterine fibroids: pooled analysis of two 12-month, placebo-controlled, randomized trials. Hum Reprod. 2019 Apr 1;34(4):623-634. doi: 10.1093/humrep/dez007. PMID 30865281
- [Derived] Larsen L, Coyne K, Chwalisz K. Validation of the menstrual pictogram in women with leiomyomata associated with heavy menstrual bleeding. Reprod Sci. 2013 Jun;20(6):680-7. doi: 10.1177/1933719112463252. Epub 2012 Nov 27. PMID 23188490